CLINICAL TRIAL: NCT02410486
Title: Early-Onset Sepsis an NICHD/CDC Surveillance Study
Acronym: EOSII
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0055; UG1HD034216 (NIH); UG1HD027904 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD027851 (NIH); UG1HD087229 (NIH); UG1HD027856 (NIH); UG1HD053109 (NIH); UG1HD068284 (NIH); UG1HD068278 (NIH); UG1HD068244 (NIH); UG1HD068263 (NIH); UG1HD027880 (NIH); UG1HD068270 (NIH); UG1HD053089 (NIH); UG1HD087226 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn, Diseases; Early Onset Neonatal Sepsis; Early-Onset Meningitis
MeSH Terms: conditions — Infant, Newborn, Diseases; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- EOS infant / mother with chorio: Infant with EOS (Gram-positive or Gram-negative) and mother with Chorioamnionitis
- EOS infant / mother without chorio: Infant with EOS (Gram-positive or Gram-negative) and mother without Chorioamnionitis
- EOS Gram-neg infant / mother with chorio: Infant with Gram-negative EOS and mother with Chorioamnionitis
- Gram-neg infant / mother without chorio: Infant with Gram-negative EOS and mother without Chorioamnionitis
- Gram-pos infant / mother with chorio: Infant with Gram-positive EOS and mother with Chorioamnionitis

SUMMARY:
This prospective surveillance study will be conducted over a 2 year period to determine current rates of Early-Onset Sepsis (EOS)/ Early-Onset Meningitis (EOM), associated pathogens, antimicrobial resistance, signs and symptoms and infant outcomes.

DETAILED DESCRIPTION:
Neonatal pathogens other than group B Streptococcus (GBS) and resistant to beta-lactam antibiotics have emerged as the most common etiologic agents of EOS and EOM among preterm and term neonates and result in high mortality rates, potentially offsetting the decreased burden of early-onset GBS disease prevented by maternal intrapartum chemoprophylaxis.

Primary Outcomes of this study:

1. To determine current hospital-based rates of early-onset neonatal infection (total, GA-specific and BW-specific, and pathogen-specific) in term and preterm infants in the era of maternal intrapartum antibiotic prophylaxis to prevent vertical transmission of group B streptococcal disease. Early-onset infection comprises EOS and/or EOM and is defined as isolation of a pathogen from blood or cerebrospinal fluid (CSF) obtained within 72 hours of birth and provision of appropriate antibiotic treatment for 5 or more days (or <5 days if death occurs while receiving antibiotic therapy).
2. To determine the antimicrobial susceptibility patterns of organisms associated with EOS and EOM

The case control aspect of this study will address 2 major conundrums regarding EOS: Can we identify risk factors for early-onset Gram-negative infections that might lead to intervention strategies to reduce risk and can we identify infants born to mothers with clinical chorioamnionitis who are at highest risk for early-onset sepsis and thus warrant antibiotic treatment soon after birth?

ELIGIBILITY:
Inclusion Criteria:

* Case Surveillance: Live born infants with gestational age of at least 22 weeks and birth weight >400 g and <72 hours of age who are delivered at NRN hospitals and have early-onset sepsis and meningitis defined as isolation of a pathogen from blood or CSF obtained within 72 hours of birth and provision of appropriate antibiotic treatment for 5 or more days (or <5 days if death occurs while receiving antibiotic therapy).
* Controls: Live born infants with gestational age of at least 22 weeks and birth weight >400 g who are delivered at NRN hospitals and have not been evaluated for early-onset sepsis (<72 hours of age) or if evaluated, they have sterile blood and/or CSF cultures and were not treated with prolonged antibiotics for clinical "culture negative" sepsis. Controls for infants with Gram-negative infection will be infants without early-onset infection. Controls for infants born to mothers with clinical chorioamnionitis will be infants without early-onset infection born to mothers with clinical chorioamnionitis. Control infants will be born at the same hospital as cases, with the same gestational age grouping as cases (22 0/7 - 28 6/7 weeks; 29 0/7 - 33 6/7 weeks; 34 0/7 - 36 6/7 weeks; and ≥ 37 weeks).

Exclusion Criteria:

* Stillbirths and infants who die in the delivery room will be excluded.
* Infants who die within 12 hours of age will be excluded if they have not been evaluated for possible infection-ie, do not have a blood culture obtained to identify EOS.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include all live born infants who are at least 22 weeks GA and have a birth weight >400 grams and are delivered at NRN centers.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine current hospital-based rates of early-onset neonatal infection | First 72 hours
To determine the antimicrobial susceptibility patterns of organisms associated with EOS and EOM | First 72 hours

SECONDARY OUTCOMES:
To identify risk factors associated with EOS/EOM due to Gram-negative pathogens (case control comparison) | First 72 hours
To determine the clinical signs/symptoms and laboratory abnormalities associated with EOS/EOM | First 72 hours
To identify risk factors for EOS/EOM in infants born to mothers with chorioamnionitis (case control comparison) | First 72 hours
To determine if term infants with EOS, identified because of maternal chorioamnionitis, can be asymptomatic at birth | First 72 hours
To determine sepsis-associated mortality rates (total, GA-specific and BW-specific, pathogen-specific) for infants with EOS/EOM | First 72 hours
To review changes over time in overall rates of EOS and EOM, pathogens associated with infection, risk factors for infection, clinical and laboratory abnormalities, and sepsis-associated mortality | 9-11 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Stoll, MD, Study Director — The University of Texas Health Science Center, Houston; Michele Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospita; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michael Cotten, MD, Principal Investigator — Duke University; Greg Sokol, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa Van Meurs, MD, Principal Investigator — Stanford University; Brenda Poindexter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kristi Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Barbara Schmidt, MD, Principal Investigator — University of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Kilpatrick R, Greenberg R, Hansen NI, Shankaran S, Carlo WA, Cotten CM, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Use and utility of C-reactive protein (CRP) in neonatal early-onset sepsis: a secondary analysis of a prospective surveillance study. J Perinatol. 2025 Jan;45(1):139-145. doi: 10.1038/s41372-024-02064-5. Epub 2024 Aug 5. PMID 39103472